CLINICAL TRIAL: NCT00659256
Title: Hepatitis C Eradication and Progression of Atherosclerosis
Brief Title: Hepatitis C Treatment and Atherosclerosis
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080106; 08-DK-0106
Record Dates: First submitted 2008-04-15; First posted 2008-04-16 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2015-03-24

CONDITIONS: Chronic Hepatitis C; Atherosclerosis
Keywords: Hepatitis C Virus; Atherosclerosis; Intima-Media Thickness; Coronary Artery Calcium Score; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Atherosclerosis; Hepatitis C

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will examine the effects of treatment for hepatitis C on atherosclerosis, or hardening of the arteries. Hepatitis C is a disease of the liver caused by a virus that can cause permanent damage to that organ. Treatment can clear the virus in at least half of patients and reduce the risk of serious complications of the disease. Atherosclerosis is an accumulation of cholesterol and fat in the arteries that can narrow blood vessels, leading to chest pain, heart attack or stroke.

Because the liver controls cholesterol and fat levels in the blood, hepatitis C infection may be a risk factor for atherosclerosis by increasing cholesterol and fat in blood vessels. Treatment of the hepatitis C may reduce the risk of atherosclerosis and its consequences. This study will determine what effect hepatitis C treatment has on the rate of atherosclerosis and narrowing of blood vessels and on the risk of heart attack or stroke.

Patients 30 years of age and older with current or past infection with hepatitis C may be eligible for this study. Participants undergo the following tests and procedures:

* Questionnaires regarding risk factors for heart disease and stroke
* Measurements of blood pressure, heart rate, weight, height, waist and hips
* Blood tests
* CT scans and ultrasound tests to measure the degree of blood vessel hardening and narrowing in the heart and neck region

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is associated with changes in lipid metabolism in the liver and the peripheral blood. Patients with chronic hepatitis C infection tend to have low levels of cholesterol and LDL-cholesterol. These levels increase in many patients after treatment and successful eradication of the virus. However, it is not known whether this increase is associated with increased cardiovascular risk and thus may increase their risk for atherosclerotic disease. To determine whether eradication of HCV affects atherosclerosis progression, we propose to examine up to 200 patients with chronic hepatitis C for markers of atherosclerosis and the risk of its complications. Up to 100 patients who have cleared HCV and recovered will be matched and compared to patients who failed to respond and continue to have chronic hepatitis C. The atherosclerosis assessment will include careful history for cardiovascular risk factors, a battery of blood tests for lipid levels and relevant biomarkers followed by specialized imaging tests of the carotid and coronary arteries, including ultrasound imaging of intima-media thickness of the carotid arteries and computerized axial tomography of the heart and coronary arteries. The primary end point in the assessment will be differences in maximal carotid intima media thickness and secondary end points will include differences in coronary artery calcium score, Framingham risk scores and other measurements or atherosclerosis. This cross-sectional study will set the stage for a more formal prospective assessment of cardiovascular risk factors and evidence of coronary and cerebrovascular disease among patients being treated with antiviral agents.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age equal to or greater than 30 years, male or female

Written informed consent

All ethnicities

Viral hepatitis status:

* Cases:

  * History of chronic hepatitis C defined by past positivity for serum HCV-RNA, HCV antibody and elevated serum alanine or aspartate aminotransferase levels for at least 6 months before start of treatment
  * Genotype 1, 2 or 3
  * Absence of detectable serum HCV-RNA by PCR on screening visit and on a previous test, at least 3 months apart. Both tests have to be performed at least 24 weeks after cessation of therapy
  * Past treatment with interferon alfa (standard or pegylated) for at least 12 weeks
  * At least 12 months after end of interferon treatment
  * Normal liver enzymes on screening visit
* Genotype 1 controls:

  * Detectable serum HCV-RNA on screening visit
  * Past treatment with interferon alfa (standard or pegylated) for at least 12 weeks
  * At least 12 months after end of interferon treatment
  * Age (difference less than or equal to 3 years), sex and race-matched with genotype 1 cases
* Genotype 2 and 3 controls:

  * Detectable serum HCV-RNA on screening visit
  * If previously treated with interferon alfa (standard or pegylated) - at least 12 months elapsed from the end of treatment
  * Age (difference less than or equal to 3 years), sex, race and genotype-matched with genotype 2 and 3 cases

EXCLUSION CRITERIA:

Pregnancy or lactation

History of clinical atherosclerotic disease manifest as:

* Ischemic cerebrovascular accident (CVA), transient ischemic accident (TIA) or radiological evidence of stroke.
* Proven coronary artery disease history of myocardial infarction, need for coronary angioplasty or coronary artery bypass graft, anginal syndrome with confirmatory stress test or cardiac imaging.
* Symptomatic peripheral vascular disease, history of angioplasty or surgical bypass.
* History of carotid artery surgery or angioplasty
* Patients with overt atherosclerotic disease can be included if the first manifestation of that disease appeared at least 3 years after cessation of interferon treatment. Control patients who were never treated in the past will not be included if there is an overt manifestation of atherosclerosis.

Diabetes mellitus unless fasting blood sugar can be maintained within normal limits and HBA1C less than 7 without the need for pharmacologic intervention

Hypertension unless blood pressures can be maintained for greater than 6 months within normal limits without the need for pharmacologic intervention

Current treatment with cholesterol lowering medications

Chronic renal failure (creatinine clearance less than 50 ml)

Known HIV infection

HCV genotype 4, 5, 6 or mixed infection.

Other causes of liver disease apart from hepatitis C (hepatitis B, alcoholic liver disease, NASH, autoimmune hepatitis, PBC etc.). Bland, non-alcoholic hepatic steatosis will not constitute an exclusion criterion

History of trauma to the neck, surgery or deformity precluding sonographic visualization of the carotid arteries

Inability to sign or understand the informed consent form

A contraindication or unwillingness to undergo the coronary calcium score CT scan will not be an exclusion criterion, as this is not a primary end-point, as long as the participant is willing to undergo an IMT measurement.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-04-08; Study Completion 2015-03-24

PRIMARY OUTCOMES:
Intima-media thickness

SECONDARY OUTCOMES:
Coronary calcium score, Framingham score

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Rotman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Maggi G, Bottelli R, Gola D, Perricone G, Posca M, Zavaglia C, Ideo G. Serum cholesterol and chronic hepatitis C. Ital J Gastroenterol. 1996 Oct-Nov;28(8):436-40. PMID 9032585
- [Background] Moriya K, Shintani Y, Fujie H, Miyoshi H, Tsutsumi T, Yotsuyanagi H, Iino S, Kimura S, Koike K. Serum lipid profile of patients with genotype 1b hepatitis C viral infection in Japan. Hepatol Res. 2003 Apr;25(4):371-376. doi: 10.1016/s1386-6346(02)00309-1. PMID 12699847
- [Background] Jarmay K, Karacsony G, Nagy A, Schaff Z. Changes in lipid metabolism in chronic hepatitis C. World J Gastroenterol. 2005 Nov 7;11(41):6422-8. doi: 10.3748/wjg.v11.i41.6422. PMID 16425410